CLINICAL TRIAL: NCT03665948
Title: The Effect of Ketogenic and Carbohydrate, Low-Glycemic Index Diet on Physical and Specific Performance Capacity, and Exercise Metabolism in Crossfit- Trained Athletes
Brief Title: Effect of Ketogenic and Carbohydrate Diet in Crossfit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Poznan University of PhysED (Individual); Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Krzysztof Durkalec-Michalski, Associate Professor, Poznan University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ULS00004
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Nutrition; Ketogenic Dieting; Low Glycemic Index Diet; Sport; Crossfit
Keywords: Sports Nutrition; Ketogenic Diet; Low Glycemic Index Diet; Crossfit; Physical capacity; Performance; Exercise metabolism; Training support

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (KD) (Experimental): Group consuming very low carbohydrate ketogenic diet. The ketogenic diet model was energetically normalized (covered the estimated energy expenditure) and assumed coverage of the daily energy requirement up to 5% of energy from carbohydrates. Proteins were administered in the amount of 1.7 g per kilogram of body mass. The remaining energy needs were covered with fats (fats covered more than 75% of the daily energy requirement). Each of the subjects in this group received 10-day menus.
  Interventions: Other: Dietary Intervention - Ketogenic Diet (KD)
- Low-Glycemic Index Diet (CHO-LGI) (Active Comparator): Group consuming carbohydrate, low-glycemic index diet. The carbohydrate diet model with a low glycemic index was energetically normalized (covered the estimated energy expenditure) and assumed coverage of the daily energy requirement of 25% of fat. Proteins were administered in the amount of 1.7 g per kilogram of body mass. The remaining energy needs were covered with carbohydrates (carbohydrates covered about ~55% of the daily energy requirement). The glycemic index of individual meals as well as the daily diet was calculated in accordance with the appropriate recommendations. Each of the subjects in this group received 10-day menus.
  Interventions: Other: Dietary Intervention - Low-Glycemic Index Diet (CHO-LGI)

INTERVENTIONS:
Other: Dietary Intervention - Ketogenic Diet (KD) — The experimental procedure for each randomly assigned participant included a 4-week of KD diet.
  Arms: Ketogenic Diet (KD)
Other: Dietary Intervention - Low-Glycemic Index Diet (CHO-LGI) — The experimental procedure for each randomly assigned participant included a 4-week of CHO-LGI diet.
  Arms: Low-Glycemic Index Diet (CHO-LGI)

SUMMARY:
The purpose of the presented study was to assess the influence of Ketogenic (KD) and a carbohydrate diet with a low glycemic index (CHO-LGI) of a 4-week diet on physical and specific performance capacity, exercise metabolism, as well as concentrations of the selected biochemical blood markers in Crossfit- trained athletes, in a randomised and parallel trial.

DETAILED DESCRIPTION:
The impact of various dietary strategies, including the alternative ketogenic diet - recently popular among strength athletes, has not been unequivocally assessed in the high-intensity sport disciplines that Crossfit belongs to. There is also a lack of data in these disciplines about the potential longer adaptation of athletes to the very low carbohydrate intake resulting from the ketogenic diet and its impact in high-intensity Crossfit training. Therefore, the purpose of this study was the assessment of the influence of a 4-week KD and a CHO-LGI diet on physical and specific performance capacity, exercise metabolism, as well as concentrations of the selected biochemical blood markers in Crossfit- trained athletes, in a randomised and parallel trial.

ELIGIBILITY:
Inclusion Criteria:

* written consent to participate,
* a current medical clearance to practice sports,
* training experience: at least 2 years,
* minimum of 4 workout sessions (Crossfit) a week.

Exclusion Criteria:

* current injury,
* any health-related contraindication,
* declared general feeling of being unwell,
* unwilling to follow the study protocol,
* smoking, illicit drug use, alcohol consumption greater than 1-2 drinks/week, dietary supplements use less than 3 weeks before the study,
* females- being pregnant or planning to become pregnant during the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Changes in aerobic capacity following dietary intervention | Baseline and after 4 weeks
Changes in CrossFit-specific performance capacity (Fight Gone Bad test) following dietary intervention | Baseline and after 4 weeks
  The number of correctly performed repetitions of exercises (reps)
Changes in energy substrates utilization following dietary intervention | Baseline and after 4 weeks
  Fats (g/min) and carbohydrates (g/min) oxidation analysis

SECONDARY OUTCOMES:
Changes in fat mass and fat free mass following dietary intervention | Baseline and after 4 weeks
  Fat mass (kg) and fat free mass (kg) analysis
Changes of red and white blood cell concentration in blood following dietary intervention | Baseline and after 4 weeks
  Red blood cells (RBC) [mln/mm³] and white blood cells (WBC) [mln/mm³] concentration analysis
Changes in blood glucose and hemoglobin concentration following dietary intervention | Baseline and after 4 weeks
  Hemoglobin (Hb) [g/dl] and glucose [g/dl] concentration analysis
Changes in blood hematocrit levels following dietary intervention | Baseline and after 4 weeks
  Hematocrit (HCT) [%] level analysis
Changes of testosterone, cortisol, urea, lactate and pyruvate concentration in blood following dietary intervention | Baseline and after 4 weeks
  Testosterone [mmol/L], cortisol [mmol/L], urea [mmol/L], lactate [mmol/L] and pyruvate [mmol/L] concentration analysis
Changes of creatine kinase, lactate dehydrogenase, alanine aminotransferase and aspartate aminotransferase activity in blood after following dietary intervention | Baseline and after 4 weeks
  Creatine kinase [U/L], lactate dehydrogenase [U/L], alanine aminotransferase [U/L] and aspartate aminotransferase [U/L] activity analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jeszka, Professor, Study Chair — Institute of Human Nutrition and Dietetics, Poznan University of Life Sciences
Locations (1):
- Institute of Human Nutrition and Dietetics, Poznan University of Life Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Shared data will be exclusively related to the level recorded indicators (anaerobic capacity and specific performance capacity indicators, exercise metabolism, levels of biochemical markers, and body composition), without personal data. The data obtained will be attached to scientific publications, depending on the requirements of the journal.

REFERENCES:
- [Derived] Durkalec-Michalski K, Nowaczyk PM, Siedzik K. Effect of a four-week ketogenic diet on exercise metabolism in CrossFit-trained athletes. J Int Soc Sports Nutr. 2019 Apr 5;16(1):16. doi: 10.1186/s12970-019-0284-9. PMID 30953522